CLINICAL TRIAL: NCT03663101
Title: A Double-blind, Randomised, Placebo Controlled, Proof-of-concept Study in Subjects With Abdominal or Thoracic Chronic Scar Pain to Assess the Analgesic Properties of Intradermal Doses of Dysport®
Brief Title: Dysport in Post-Surgical Neuralgia
Acronym: PMOD03
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D-FR-52120-244; 2018-001703-37 (EudraCT Number)
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Results first posted 2020-12-04 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Chronic Scar Pain
MeSH Terms: interventions — Lidocaine; Botulinum Toxins, Type A; abobotulinumtoxinA; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Pre-Randomization, Run-In period (part A) (Experimental): Crossover run-in part A - Subjects will be injected (Test 1) with either saline or local anaesthetic (lidocaine). One week later, they will be crossed over, injected with the other agent (Test 2).
  Interventions: Drug: Lidocaine; Drug: Placebo
- Dysport dose 1 (part B) (Experimental): Dysport dose 1 as a single-dose, intradermal injection.
  Interventions: Biological: Botulinum toxin type A
- Dysport dose 2 (part B) (Experimental): Dysport dose 2 as a single-dose, intradermal injection.
  Interventions: Biological: Botulinum toxin type A
- Dysport dose 3 (part B) (Experimental): Dysport dose 3 as a single-dose, intradermal injection.
  Interventions: Biological: Botulinum toxin type A
- Placebo (saline solution) (part B) (Placebo Comparator): Placebo single-dose, intradermal injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — 0.5 mL (2.5 mg) of lidocaine per injection point will be injected subcutaneously (maximum 10 injection points).
  Arms: Pre-Randomization, Run-In period (part A)
Biological: Botulinum toxin type A — 0.2 mL of one of three different doses of Dysport per injection point will be injected intradermally (maximum 10 injection points).
  Other Names: AbobotulinumtoxinA (Dysport®)
  Arms: Dysport dose 1 (part B); Dysport dose 2 (part B); Dysport dose 3 (part B)
Drug: Placebo — Part A - 0.5 mL of sodium chloride solution 0.9% (saline solution) per injection point will be injected subcutaneously (maximum 10 injection points).
  Other Names: Saline solution
  Arms: Pre-Randomization, Run-In period (part A)
Drug: Placebo — Part B - 0.2 mL of sodium chloride solution 0.9% (saline solution) per injection point will be injected intradermally (maximum 10 injection points, 2,0 mL maximum).
  Arms: Placebo (saline solution) (part B)

SUMMARY:
The study is designed to determine whether a currently licensed version of botulinum toxin (Dysport®) is effective for the treatment of pain that has developed and/or persisted for months or years around the scar of a previous surgical site, and whether this condition could be suitable for the testing of similar new medicines. The study will compare three different doses of Dysport® to see if there is benefit and/or a best dose for treating persistent post-surgery scar pain.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged between 18 and 75 years inclusive at the time of giving informed consent.
* Subjects suffering from an area of chronic pain post-abdominal or thoracic surgery, chronic abdominal or thoracic scar pain.
* Longitudinal axis of the pain area of 10 cm long maximum (as mapped upon screening).
* Subjects with moderate to severe pain, i.e. spontaneous NRS score of 4-8 which has been stable for the previous month before screening.
* Stable use of analgesics (or any medication impacting pain perception) during the month before screening and expected to be stable for the study duration.
* Under stable medication regimen for other medication, i.e. during the month before screening.
* Time from surgery which caused the painful scar more than six months and less than ten years at screening.
* No other distracting pain either chronic or acute.
* Female subjects of childbearing potential must have a negative urine pregnancy test result and be willing to use reliable contraceptive measures throughout study participation.
* The subject's primary care physician has provided evidence which can be used to confirm that within the last 12 months of dosing that there is nothing in their medical history that would preclude their enrolment into a clinical study.

Exclusion Criteria:

* Previous treatment with Botulinum neurotoxin (BTX) (any serotype) during the past six months before screening.
* History of hypersensitivity to any of the components of the Dysport formulation (which includes human serum albumin and lactose) or allergy to cow's milk protein.
* Known hypersensitivity to lidocaine or other anaesthetics of the amide type, known hypersensitivity to hydroxybenzoates, complete heart block, hypovolaemia.
* Any medical condition that may put the subject at risk with exposure to BTX, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other disease that might interfere with neuromuscular function.
* Opioid analgesic use at a Morphine Equivalent Dosage (MED) of >75mg per day.
* Neuroma in the scar pain area, diagnosed per ultrasound.
* Use of agents that could interfere with neuromuscular transmission, including calcium channel blockers, penicillamine, aminoglycosides, lincosamides, polymixins, magnesium sulphate, anticholinesterases, succinylcholine and quinidine.
* Need of any prohibited medication.
* Any abnormal laboratory value, physical examination, vital signs, or electrocardiogram (ECG) that, in the opinion of the investigator, is clinically significant and that would compromise the safety of the subject in the study.
* Positive for hepatitis B antigen or hepatitis C virus ribonucleic acid, positive results for human immunodeficiency virus, or who receives diagnosis for acquired immunodeficiency syndrome.
* Positive urine screen for drugs of abuse (except for cotinine and unless explained by the investigator for therapeutic use of medication) or any history of drug or alcohol abuse, misuse, physical or psychological dependence, mood changes, sleep disturbance and functional capacity which have an impact on pain perception.
* Significant neurological or psychiatric disorders including mental instability (unrelated to the pain) that could interfere with pain assessments; other pre-existing pain syndromes, acute or chronic, that might impair the assessment of the scar pain.
* Any medical history of significance and/or inadequately controlled such as cardiovascular (e.g. uncontrolled high blood pressure, high risk of cardiovascular events, severe heart failure), pulmonary (e.g. uncontrolled asthma or emphysema), haematologic, (e.g. coagulopathy/bleeding disorders), neurological (e.g. swallowing problems, blurred or double vision, trouble saying words clearly (dysarthria), hoarseness or change or loss of voice (dysphonia)), liver disease (e.g. severe hepatic impairment), kidney disease (e.g. impaired renal function in subjects taking diuretics, angiotensin converting enzyme (ACE)-inhibitors, or angiotensin II antagonists), endocrine, immunologic, dermatologic painful conditions or any other conditions that may compromise in the opinion of the investigator the ability of the subject to participate in the study.
* Subjects who participated in a clinical research study involving a new chemical entity or an experimental drug within 30 days before screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- St Pancras Clinical Research, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase II proof-of-concept study was conducted at single investigational site in the United Kingdom between 30 October 2018 and 08 November 2019. The study consisted of two sequential parts: Part A (Pre-randomisation run-in period) and Part B (Randomised double-blind period). Part A was considered as an extended screening period.
Pre-assignment Details: Part A was conducted to identify participants who would potentially benefit from Dysport® injection, considered as 'responders'. Part B was a double-blind study of Dysport or placebo injection in responders from Part A. Of the 46 participants who were included in Part A, 17 were responders. Of which, 16 participants were randomised into Part B of the study.
Groups:
- Placebo: Participants received a single dose of placebo (matching with Dysport) intradermal injection per injection point (maximum of 10 injection points) on Day 1. Injections were performed under a constant volume of 0.2 milliliters (mL).
- Dysport 2.5 U/Injection Site: Participants received a single dose of Dysport 2.5 units (U) intradermal injection per injection point (maximum of 10 injection points) on Day 1. The maximal total dose was 25 U. Injections were performed under a constant volume of 0.2 mL.
- Dysport 10 U/Injection Site: Participants received a single dose of Dysport 10 U intradermal injection per injection point (maximum of 10 injection points) on Day 1. The maximal total dose was 100 U. Injections were performed under a constant volume of 0.2 mL.
- Dysport 20 U/Injection Site: Participants received a single dose of Dysport 20 U intradermal injection per injection point (maximum of 10 injection points) on Day 1. The maximal total dose was 200 U. Injections were performed under a constant volume of 0.2 mL.
Period: Overall Study
Arm/Group | Placebo | Dysport 2.5 U/Injection Site | Dysport 10 U/Injection Site | Dysport 20 U/Injection Site
Started | 4 | 3 | 5 | 4
Completed | 4 | 3 | 5 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomised population included all participants randomised in the double-blind period (Part B).
Groups:
- Placebo: Participants received a single dose of placebo (matching with Dysport) intradermal injection per injection point (maximum of 10 injection points) on Day 1. Injections were performed under a constant volume of 0.2 mL.
- Dysport 2.5 U/Injection Site: Participants received a single dose of Dysport 2.5 U intradermal injection per injection point (maximum of 10 injection points) on Day 1. The maximal total dose was 25 U. Injections were performed under a constant volume of 0.2 mL.
- Total: Total of all reporting groups
Arm/Group | Placebo | Dysport 2.5 U/Injection Site | Dysport 10 U/Injection Site | Dysport 20 U/Injection Site | Total
Number analyzed (Participants) | 4 | 3 | 5 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (10.7) | 49.7 (6.0) | 46.0 (11.3) | 48.8 (16.7) | 50.0 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 2 | 11
  Male | 1 | 0 | 2 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 4 | 3 | 2 | 3 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Onset of Effect in the Spontaneous Numerical Rating Scale (NRS) Score
Description: The time to onset of effect was defined as the time to a decrease from baseline of two points or greater in the spontaneous NRS score. Pain intensity was scored using an 11-point NRS score ranging from 0 to 10, where 0= no pain and 10= worst possible pain. Participants were provided with an Actiwatch® during an Actiwatch® training visit to record their spontaneous NRS scores at home. The Actiwatch® alerted the participants twice a day to record their average and maximal NRS scores over the preceding 12 hours. The questions were asked of the participants by the Actiwatch®: "Please rate your pain by selecting the one number that best describes your pain on average during the last 12 hours." and "Please rate your pain by selecting the one number that best describes your pain at its worst during the last 12 hours." Only descriptive statistical analysis was performed for this outcome measure.
Time Frame: Part B: From baseline (defined as mean of all predose data from Day -7 and including predose on Day 1) up to end of study (Week 16) or early discontinuation.
Population: Randomised population included all participants randomised in the double-blind period (Part B). Only participants who reached the time to onset were analysed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Dysport 2.5 U/Injection Site | Dysport 10 U/Injection Site | Dysport 20 U/Injection Site
Number analyzed (Participants) | 4 | 3 | 5 | 4
days
  Worst NRS score: number analyzed (Participants) | 2 | 3 | 5 | 2
  Worst NRS score | 4.41 (4.92) | 15.11 (25.17) | 29.45 (39.82) | 0.65 (0.32)
  Average NRS score: number analyzed (Participants) | 3 | 3 | 4 | 2
  Average NRS score | 6.75 (2.74) | 31.63 (53.78) | 4.60 (6.55) | 0.90 (0.03)

2. Primary Outcome: Peak Effect in the Spontaneous NRS Score
Description: The peak effect was defined as the maximal decrease from baseline in the spontaneous NRS score over a 12-hour period. Pain intensity was scored using an 11-point NRS score ranging from 0 to 10, where 0= no pain and 10= worst possible pain. Participants were provided with an Actiwatch® during an Actiwatch® training visit to record their spontaneous NRS scores at home. The Actiwatch® alerted the participants twice a day to record their average and maximal NRS scores over the preceding 12 hours. The questions were asked of the participants by the Actiwatch®: "Please rate your pain by selecting the one number that best describes your pain on average during the last 12 hours." and "Please rate your pain by selecting the one number that best describes your pain at its worst during the last 12 hours." Greater reductions in change from baseline correspond to greater pain relief.
Time Frame: as for outcome 1
Population: Randomised population included all participants randomised in the double-blind period (Part B).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Dysport 2.5 U/Injection Site | Dysport 10 U/Injection Site | Dysport 20 U/Injection Site
Number analyzed (Participants) | 4 | 3 | 5 | 4
score on a scale
  Worst NRS score | -2.36 (1.58) | -4.73 (0.55) | -3.54 (2.15) | -2.82 (2.91)
  Average NRS score | -2.52 (0.91) | -3.53 (0.45) | -3.72 (1.57) | -2.12 (2.37)

3. Primary Outcome: Time to Peak Effect in the Spontaneous NRS Score
Description: The time to peak effect was defined as the time to reach the peak effect over a 12-hour period. Pain intensity was scored using an 11-point NRS score ranging from 0 to 10, where 0= no pain and 10= worst possible pain. Participants were provided with an Actiwatch® during an Actiwatch® training visit to record their spontaneous NRS scores at home. The Actiwatch® alerted the participants twice a day to record their average and maximal NRS scores over the preceding 12 hours. The questions were asked of the participants by the Actiwatch®: "Please rate your pain by selecting the one number that best describes your pain on average during the last 12 hours." and "Please rate your pain by selecting the one number that best describes your pain at its worst during the last 12 hours."
Time Frame: as for outcome 1
Population: Randomised population included all participants randomised in the double-blind period (Part B).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Dysport 2.5 U/Injection Site | Dysport 10 U/Injection Site | Dysport 20 U/Injection Site
Number analyzed (Participants) | 4 | 3 | 5 | 4
days
  Worst NRS score | 10.63 (10.18) | 33.46 (51.41) | 41.94 (35.72) | 3.11 (1.56)
  Average NRS score | 12.51 (7.26) | 33.13 (52.51) | 11.04 (11.58) | 26.49 (49.89)

4. Primary Outcome: Duration of Effect in the Spontaneous NRS Score
Description: The duration of effect was defined as the duration between time to onset and last timepoint for which decrease from baseline in the spontaneous NRS score was two points or greater. Pain intensity was scored using an 11-point NRS score ranging from 0 to 10, where 0= no pain and 10= worst possible pain. Participants were provided with an Actiwatch® during an Actiwatch® training visit to record their spontaneous NRS scores at home. The Actiwatch® alerted the participants twice a day to record their average and maximal NRS scores over the preceding 12 hours. The questions were asked of the participants by the Actiwatch®: "Please rate your pain by selecting the one number that best describes your pain on average during the last 12 hours." and "Please rate your pain by selecting the one number that best describes your pain at its worst during the last 12 hours."
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Dysport 2.5 U/Injection Site | Dysport 10 U/Injection Site | Dysport 20 U/Injection Site
Number analyzed (Participants) | 4 | 3 | 5 | 4
days
  Worst NRS score: number analyzed (Participants) | 2 | 3 | 5 | 2
  Worst NRS score | 86.04 (25.52) | 86.68 (23.89) | 66.80 (44.28) | 110.52 (0.74)
  Average NRS score: number analyzed (Participants) | 3 | 3 | 4 | 2
  Average NRS score | 53.53 (51.44) | 65.17 (58.21) | 102.75 (18.36) | 110.02 (1.45)

5. Secondary Outcome: Change From Baseline in the Spontaneous NRS Score Throughout the Study
Description: Pain intensity was scored using an 11-point NRS score ranging from 0 to 10, where 0= no pain and 10= worst possible pain. Participants were provided with an Actiwatch® during an Actiwatch® training visit to record their spontaneous NRS scores at home. The Actiwatch® alerted the participants twice a day to record their average and maximal NRS scores over the preceding 12 hours. The questions were asked of the participants by the Actiwatch®: "Please rate your pain by selecting the one number that best describes your pain on average during the last 12 hours." and "Please rate your pain by selecting the one number that best describes your pain at its worst during the last 12 hours." Greater reductions in change from baseline correspond to greater pain relief.
Time Frame: as for outcome 1
Population: Randomised population included all participants randomised in the double-blind period (Part B).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Dysport 2.5 U/Injection Site | Dysport 10 U/Injection Site | Dysport 20 U/Injection Site
Number analyzed (Participants) | 4 | 3 | 5 | 4
score on a scale
  Daily worst NRS score: Baseline | 5.1 (1.0) | 5.1 (1.0) | 5.3 (1.6) | 5.8 (0.9)
  Daily worst NRS score: Week 2: number analyzed (Participants) | 4 | 3 | 4 | 4
  Daily worst NRS score: Week 2 | -0.6 (0.9) | -2.1 (2.1) | -1.4 (3.5) | -1.1 (2.7)
  Daily worst NRS score: Week 4: number analyzed (Participants) | 4 | 3 | 4 | 4
  Daily worst NRS score: Week 4 | -1.6 (1.8) | -2.1 (1.8) | -1.4 (4.2) | -1.6 (2.7)
  Daily worst NRS score: Week 6: number analyzed (Participants) | 4 | 3 | 4 | 4
  Daily worst NRS score: Week 6 | -1.1 (0.7) | -0.1 (1.0) | -1.7 (2.9) | -1.6 (2.6)
  Daily worst NRS score: Week 12: number analyzed (Participants) | 3 | 3 | 5 | 4
  Daily worst NRS score: Week 12 | -0.5 (1.4) | -1.4 (0.6) | -0.7 (1.1) | -0.8 (3.3)
  Daily worst NRS score: Week 16: number analyzed (Participants) | 3 | 3 | 5 | 4
  Daily worst NRS score: Week 16 | -0.0 (2.0) | -1.4 (1.1) | -1.3 (3.1) | -0.3 (1.7)
  Daily average NRS score: Baseline | 4.5 (1.1) | 3.9 (1.0) | 4.7 (1.2) | 4.9 (1.2)
  Daily average NRS score: Week 2: number analyzed (Participants) | 4 | 3 | 4 | 4
  Daily average NRS score: Week 2 | -0.9 (1.0) | -2.0 (1.8) | -2.1 (2.8) | -1.7 (2.5)
  Daily average NRS score: Week 4: number analyzed (Participants) | 4 | 3 | 4 | 4
  Daily average NRS score: Week 4 | -1.6 (1.9) | -1.9 (1.3) | -2.1 (3.2) | -1.4 (2.0)
  Daily average NRS score: Week 6: number analyzed (Participants) | 4 | 3 | 4 | 4
  Daily average NRS score: Week 6 | -1.0 (0.9) | -0.4 (2.0) | -2.0 (2.6) | -1.4 (2.0)
  Daily average NRS score: Week 12: number analyzed (Participants) | 3 | 3 | 5 | 4
  Daily average NRS score: Week 12 | -0.5 (1.6) | -1.5 (0.6) | -1.2 (1.9) | -0.6 (2.5)
  Daily average NRS score: Week 16: number analyzed (Participants) | 3 | 3 | 5 | 4
  Daily average NRS score: Week 16 | -0.6 (1.5) | -0.9 (0.8) | -1.6 (2.3) | -0.4 (1.5)

6. Secondary Outcome: Change From Baseline in the Stimulus-Evoked NRS Score on the Painful Area at Weeks 6 and 12
Description: For stimulus-evoked NRS score during Quantitative Sensory Testing, participants were submitted to stimuli of various nature (light touch, pressure and temperature) applied to the painful area. Pain intensity was scored using an 11-point NRS score ranging from 0 to 10, where 0= no pain and 10= worst possible pain. Static mechanical allodynia is the response to light sustained normally innocuous pressure against the skin. Dynamic mechanical allodynia is the response to a normally innocuous light moving mechanical stimulus on the skin. Temporal summation is a condition, which demonstrates an increased perception of pain to repetitive painful stimuli.
Time Frame: Part B: Baseline (defined as mean of all predose data from Day -7 and including predose on Day 1) and Weeks 6 and 12
Population: Randomised population included all participants randomised in the double-blind period (Part B).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Dysport 2.5 U/Injection Site | Dysport 10 U/Injection Site | Dysport 20 U/Injection Site
Number analyzed (Participants) | 4 | 3 | 5 | 4
score on a scale
  Static mechanical allodynia: Baseline | 1.3 (1.5) | 3.0 (3.6) | 4.2 (1.1) | 4.5 (3.1)
  Static mechanical allodynia: Week 6 | 1.0 (1.2) | -1.7 (4.0) | -2.6 (1.8) | -1.0 (5.5)
  Static mechanical allodynia: Week 12 | 0.8 (1.0) | -0.3 (5.7) | -2.0 (1.4) | -0.8 (5.1)
  Dynamic mechanical allodynia: Baseline | 1.3 (1.0) | 2.3 (3.2) | 2.4 (1.7) | 5.3 (1.0)
  Dynamic mechanical allodynia: Week 6 | -0.5 (1.0) | -1.7 (2.1) | -2.0 (1.9) | -2.5 (2.6)
  Dynamic mechanical allodynia: Week 12 | -0.3 (2.1) | -1.3 (1.5) | -0.2 (1.5) | -2.0 (2.7)
  Temporal summation: Baseline | 1.5 (1.3) | 0.3 (1.5) | 3.6 (3.0) | 1.8 (2.1)
  Temporal summation: Week 6 | 1.8 (2.1) | 0.3 (0.6) | 1.8 (1.1) | 2.8 (1.7)
  Temporal summation: Week 12 | 2.0 (0.8) | 0.3 (3.1) | 1.4 (1.1) | 2.8 (1.7)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the start of study drug administration (Day 1) in Part B up to end of study visit or early discontinuation, approximately 16 weeks.
Description: Safety population included all participants who received at least one dose of the study drug during the randomised double-blind period (Part B).
Arm/Group | Placebo | Dysport 2.5 U/Injection Site | Dysport 10 U/Injection Site | Dysport 20 U/Injection Site
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/3 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 3/4 | 3/3 | 4/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | Dysport 2.5 U/Injection Site (N=3) | Dysport 10 U/Injection Site (N=5) | Dysport 20 U/Injection Site (N=4)
Pancreatogenous diabetes (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | Dysport 2.5 U/Injection Site (N=3) | Dysport 10 U/Injection Site (N=5) | Dysport 20 U/Injection Site (N=4)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hyporeflexia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensory loss (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric mucosa erythema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic failure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site rash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hereditary non-polyposis colorectal cancer syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device physical property issue (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Recruitment was closed prematurely by 30 June 2019 due to slow enrolment (16 participants randomized instead of 24 initially planned), which meant Sponsor did not believe it was feasible to continue study in an acceptable timeframe. The decision was not related to any safety/tolerability concern with Dysport.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT03663101/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-28): https://cdn.clinicaltrials.gov/large-docs/01/NCT03663101/SAP_001.pdf